CLINICAL TRIAL: NCT06021964
Title: Prospective Cohort Observational Study of Placenta Accreta Spectrum Disorders
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Guangzhou Medical University (Other)
Collaborators: Peking University Third Hospital (Other); Department of Obstetrics and Gynecology, Nanfang Hospital, Southern Medical University (Unknown); Peking Union Medical College Hospital (Other); TONGJI MEDICAL COLLEGE OF HUST (Unknown); First Affiliated Hospital of Chongqing Medical University (Other); West China Second University Hospital,Sichuan University / West China women's and children's Hospital (Unknown); Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dunjin Chen, Department of Gynecology and Obstetrics, the Third Affiliated Hospital of Guangzhou Medical University, Guangzhou Medical University
Other Study IDs: 2022YFC2704501
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Placenta Accreta Spectrum Disorders,Previous Cesarean Section
Keywords: placenta accreta spectrum disorders；Previous cesarean section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The incidence of placenta accreta spectrum disorders has shown an increasing trend worldwide due to the increase of cesarean section rate. Research on the outcomes of placenta accreta spectrum disorders primarily relies on retrospective analysis. The aim of this study was to establish a prospective, multicenter cohort in China in order to conduct further investigations on the clinical features, predictive capabilities, diagnostic methods, and pathogenesis of placenta accreta spectrum disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women aged 18-45;
2. at least one previous cesarean section ,regular antenatal examination and plan to give birth at research center
3. sign informed consent

Exclusion Criteria:

Irregular antenatal examination; Twins; Autoimmune diseases; Prepregnancy hypertension; Prepregnancy diabetes mellitus; Inheritance Sexual diseases; tumor; Abnormal liver and kidney function in early pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women aged 18-45 who at least had one previous cesarean section
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-28 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of placenta accreta spectrum disorders | baseline

SECONDARY OUTCOMES:
Preterm delivery Preterm delivery | baseline
Blood lost during delivery | baseline
Blood loss in the first 24 hours of delivery | baseline
hysterectomy | baseline
Blood transfusion | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Key Laboratory for Major Obstetric Diseases of Guangdong Province, Guangdong Provincial Clinical Research Center for Obstetrics and Gynecology，The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided